CLINICAL TRIAL: NCT03371485
Title: A Cancer Research UK Phase I Trial of AST-VAC2 (Allogeneic Dendritic Cell Vaccine) Administered Weekly Via Intradermal Injection in Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: AST-VAC2 Vaccine in Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/17/003; 2016-002577-35 (EudraCT Number)
Record Dates: First submitted 2017-09-29; First posted 2017-12-13 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-03

CONDITIONS: Advanced Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Immunotherapy; Cancer vaccine; Dendritic cell vaccine; Allogeneic vaccine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with advanced NSCLC, to receive AST-VAC2 (Experimental): Participants will receive up to a maximum of six vaccinations over six weeks. Each weekly AST-VAC2 vaccination will be administered as a split dose via two intradermal injections at a target dose defined as 1 x 10^7 viable cells. There is no dose escalation planned during the study; only one dose level will be explored.
  Interventions: Biological: AST-VAC2

INTERVENTIONS:
Biological: AST-VAC2 — Allogeneic dendritic cell vaccine.

SUMMARY:
This clinical study is looking at a vaccine called AST-VAC2 in adult patients with advanced non-small cell lung cancer (NSCLC). The main aim of the study: If the dose can be given safely to patients, learn more about the potential side effects of the vaccine and how they can be managed and also what happens to AST-VAC2 inside the body.

DETAILED DESCRIPTION:
This clinical study is looking at a vaccine called AST-VAC2. AST-VAC2 has been designed to potentially help the immune system attack the cancer. This is a new vaccine which looks promising in laboratory studies but it has never been tested in man.

Dendritic cells occur naturally in your body as part of the immune system however these dendritic cells have a special role in finding proteins in the body which are associated with cancer and it is hoped that the vaccine will train the immune system to recognise these proteins and attack the cancer.

Some cancers tend to have more of a certain type of protein (part of the body's building blocks that make up cells) called 'hTERT' and it has been shown in laboratory studies (and also studies in patients using a similar type of vaccine), that targeting hTERT can lead to destruction of cancer cells by the immune system. AST-VAC2 will target the hTERT protein.

Human Leukocyte Antigen (HLA) is another type of protein. An HLA pre-screening test will be able to show if a person is positive or negative for a specific HLA protein (AST-VAC2 can only work with some types of HLA), as being positive for the protein may mean there is a better chance of the vaccine attacking the cancer. Patients who are positive for the specific HLA type will be asked to consent to the vaccine. Those patients who are negative for the HLA type will not be eligible for the trial.

ELIGIBILITY:
Inclusion Criteria:

1. a) Patients with advanced NSCLC (metastatic or locally advanced), for whom there are no other suitable treatment options.-

   * Able to and likely to be well enough to receive six vaccinations i.e. judged by the Investigator to not require alternate treatment for the duration of the vaccination schedule and period to end of vaccination visit.
   * Has had sufficient wash out periods from previous treatments as follows:

     i) four weeks for chemotherapy ii) six weeks for investigational medicinal products (IMPs) iii) eight weeks for immunotherapy (shorter intervals may be acceptable based on half-life of treatment. Eligibility will be confirmed by the Sponsor and CI).
   * Measurable disease
   * Biopsiable disease is preferable however patients without biopsiable disease can still be considered for the study.
2. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up.
3. Confirmed HLA A*02:01 positive genotype.
4. Life expectancy of at least 12 weeks.
5. World Health Organisation (WHO) performance status of 0-2.
6. Haematological and biochemical indices within the ranges shown below. These measurements must be performed prior to the patient receiving the first AST-VAC2 vaccination.

   Laboratory Test and Value required

   Haemoglobin (Hb) ≥9.0 g/dL; Absolute neutrophil count (ANC) ≥1.5 x 10^9 /L; Platelet count ≥100 x 10 ^9/L; Lymphocyte count ≥1.0 x 10^9 /L; Bilirubin ≤1.5 x upper limit of normal (ULN); Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) and alkaline phosphatase (ALP) ≤ 3.0 x ULN; Calculated creatinine clearance > 30 mL/min
7. 18 years or over at the time consent is given.

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons) during the previous four weeks before treatment.
2. Ongoing toxic manifestations of previous treatments greater than CTCAE Grade 1. Exceptions to this are alopecia or certain Grade 2 toxicities, which in the opinion of the Investigator and the Sponsor should not exclude the patient.
3. Systemic steroids or other drugs with a likely effect on immune competence are forbidden during the trial with the exception of replacement treatment. Inhaled and topical steroids are permitted. The predictable need of their use will preclude the patient from trial entry.
4. Female patients who are able to become pregnant (or are already pregnant or lactating). However, those patients who have a negative serum or urine pregnancy test before enrolment and agree to use two forms of contraception (one effective form plus a barrier method) [oral, injected or implanted hormonal contraception and condom; intra-uterine device and condom; diaphragm with spermicidal gel and condom] or agree to sexual abstinence*, effective from the first administration of AST-VAC2 throughout the trial and for six months afterwards are considered eligible.
5. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using a barrier method of contraception [condom plus spermicide] or to sexual abstinence* effective from the first administration of AST-VAC2, throughout the trial and for six months afterwards. Men with partners of child-bearing potential must also be willing to ensure that their partner uses an effective method of contraception for the same duration for example, hormonal contraception, intrauterine device, diaphragm with spermicidal gel or sexual abstinence). Men with pregnant or lactating partners must be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure of the foetus or neonate.

   *Abstinence is only considered to be an acceptable method of contraception when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
6. Major thoracic or abdominal surgery from which the patient has not yet recovered.
7. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
8. Known to be serologically positive for Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV).
9. Evidence of any ongoing active autoimmune disease.
10. Concurrent congestive heart failure, prior history of class III/ IV cardiac disease (New York Heart Association [NYHA]), prior history of cardiac ischaemia or prior history of cardiac arrhythmia.
11. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I trial of AST-VAC2. Participation in an observational trial or interventional clinical trial which does not involve administration of an IMP and which would not place an unacceptable burden on the patient in the opinion of the Investigator and Medical Advisor would be acceptable.
12. Any vaccination given within four weeks before the first AST-VAC2 vaccination (except for COVID-19 vaccinations which are permitted at investigators discretion).
13. Any planned prophylactic vaccination from trial entry until completion of the AST-VAC2 vaccinations (except for COVID-19 vaccinations which are permitted at investigators discretion).
14. Any condition which might interfere with the patient's ability to generate an immune response.
15. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Middleton, Prof, Principal Investigator — The Queen Elizabeth Hospital
Locations (2):
- United Kingdom (2):
  - Queen Elizabeth Hospital, Birmingham
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Simple summary of trial on Cancer Research UK website. — https://www.cancerresearchuk.org/about-cancer/find-a-clinical-trial/a-trial-of-a-vaccine-called-ast-vac2-for-non-small-cell-lung-cancer

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial participants were enrolled at two trial sites between 29 May 2018 and 04 February 2022.
Period: Main Trial (6 AST-VAC2 Vaccinations)
Arm/Group | Participants With Advanced NSCLC, to Receive AST-VAC2
Started | 9
Completed | 8
Not Completed | 1
Not completed — Participant died before receiving AST-VAC2. | 1
Period: 2-year Follow-up
Arm/Group | Participants With Advanced NSCLC, to Receive AST-VAC2
Started | 8
Completed | 3
Not Completed | 5
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Advanced NSCLC, to Receive AST-VAC2
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 56 [53 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9

OUTCOME MEASURES:

1. Primary Outcome: Frequency and Causality of Serious Adverse Events (SAEs), Non-Serious Adverse Events (NSAEs) and Grade ≥3 Adverse Events (AEs) to AST-VAC2
Description: Number of SAEs, NSAEs and Grade ≥3 AEs overall and number of SAEs, NSAEs and Grade ≥3 AEs related to AST-VAC2. AEs categorised according to Medical Dictionary for Regulatory Activities (MedDRA) version (v) 25.0 and graded for severity according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.02 or protocol specific grading system for injection site reactions (ISRs; Section 9.8 of protocol). AEs assessed by the reporting study doctors for a causal relationship to AST-VAC2. Related are those AEs with a causality of possible, probable or highly probable. All AEs and SAEs were collected until 30 days post last vaccination but only related AEs and SAEs were collected thereafter.
Time Frame: From the time of informed consent up to 2 years from the first dose of AST-VAC2, a median (range) of 402.5 days (101-770).
Population: Safety Population: All enrolled participants who received at least one AST-VAC2 vaccination. This population will also be used for overall survival at 2 years post first AST-VAC2 vaccination. Participants are evaluable for survival regardless of whether they go on to receive another anti-cancer therapy.
Measure: Number; unit: Adverse Events
Arm/Group | Participants With Advanced NSCLC, to Receive AST-VAC2
Number analyzed (Participants) | 8
Adverse Events
  Total SAEs | 0
  Total NSAEs | 97
  Grade ≥3 AEs | 3
  Related SAEs | 0
  Related NSAEs | 59
  Related Grade ≥3 AEs | 1

2. Primary Outcome: Number of Participants Experiencing ISRs by Grade
Description: Number of participants experiencing ISRs Grade 1 to 4 according to protocol-specific grading of ISRs (protocol section 9.8); Grade 1: minimal effect on activities of daily living, Grade 2: restricts activities of daily living, Grade 3: prevents/severely limits activities of daily living, Grade 4: life-threatening consequences; urgent intervention indicated. Participants may have had ISRs of different grades at different vaccinations and are counted once for each grade of ISR reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Advanced NSCLC, to Receive AST-VAC2
Number analyzed (Participants) | 8
Participants
  Total Grade 1 ISRs | 8
  Total Grade 2 ISRs | 2
  Total Grade 3 ISRs | 0
  Total Grade 4 ISRs | 0

3. Secondary Outcome: Number of Participants Showing a Durable Peripheral Immune Response
Description: Immunological response in whole blood (peripheral blood mononuclear cells) by human telomerase reverse transcriptase (hTERT) specific T cells measured by enzyme-linked immunospot (ELISPOT), with a durable peripheral immune response defined as a change in one validated assay at two time points after at least two vaccinations (where a change is defined as 2.5 fold change over baseline [after removal of background], assay control and >35 spots/10^6 cells).
Time Frame: Screening, vaccination weeks 3, 4 and 6; 2 weeks post last vaccination and 3, 6 and 12 months post first vaccination.
Population: Secondary Immunogenicity Endpoint Population: All eligible participants who received at least 3 AST-VAC2 vaccinations and had baseline and at least 2 post-vaccination blood samples taken.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Advanced NSCLC, to Receive AST-VAC2
Number analyzed (Participants) | 8
Participants | 2

4. Secondary Outcome: Mean Fold Change in hTERT Specific T Cells Over Baseline by Timepoint: hTERT Peptide Pool 1 Assay (p1-387)
Description: Immunological response in whole blood (peripheral blood mononuclear cells) by hTERT specific T cells measured by ELISPOT and presented as mean fold change in spots/10^6 cells (after removal of background) from baseline to each timepoint assessed. Mean (full range) data are reportable data from the participants analysed at each timepoint. Non-reportable data and timepoints where no participants had reportable data are not shown.
Time Frame: Screening, vaccination weeks 3, 4 and 6; 2 weeks post last vaccination and 3, 6 and 12 months post first vaccination.
Population: Secondary Immunogenicity Endpoint Population: All eligible participants who received at least 3 AST-VAC2 vaccinations and had baseline and at least 2 post-vaccination blood samples taken (N=8). Some participants did not have data at all timepoints.
Measure: Mean (Full Range); unit: Fold Change from Baseline
Arm/Group | Participants With Advanced NSCLC, to Receive AST-VAC2
Number analyzed (Participants) | 8
Fold Change from Baseline
  Week 3 Vaccination: number analyzed (Participants) | 6
  Week 3 Vaccination | 29.54 [29.54 to 29.54]
  3 months post first vaccination: number analyzed (Participants) | 4
  3 months post first vaccination | 29.75 [29.75 to 29.75]

5. Secondary Outcome: Mean Fold Change in hTERT Specific T Cells Over Baseline by Timepoint: hTERT Peptide Pool 2 Assay (p377-763)
Description: as for outcome 4
Time Frame: Screening, vaccination weeks 3, 4 and 6; 2 weeks post last vaccination and 3, 6 and 12 months post first vaccination.
Population: as for outcome 4
Measure: Mean (Full Range); unit: Fold Change from Baseline
Arm/Group | Participants With Advanced NSCLC, to Receive AST-VAC2
Number analyzed (Participants) | 8
Fold Change from Baseline
  Week 3 Vaccination: number analyzed (Participants) | 6
  Week 3 Vaccination | 156.89 [30.10 to 283.67]
  Week 4 Vaccination: number analyzed (Participants) | 5
  Week 4 Vaccination | 118.78 [32.55 to 205.00]
  Week 6 Vaccination | 47.90 [47.90 to 47.90]
  2 weeks post last vaccination: number analyzed (Participants) | 4
  2 weeks post last vaccination | 269.00 [269.00 to 269.00]
  3 months post first vaccination: number analyzed (Participants) | 4
  3 months post first vaccination | 331.67 [331.67 to 331.67]
  6 months post first vaccination: number analyzed (Participants) | 3
  6 months post first vaccination | 331.00 [331.00 to 331.00]
  12 months post first vaccination: number analyzed (Participants) | 2
  12 months post first vaccination | 72.60 [72.60 to 72.60]

6. Secondary Outcome: Mean Fold Change in hTERT Specific T Cells Over Baseline by Timepoint: hTERT Peptide Pool 3 Assay (p753-1132)
Description: as for outcome 4
Time Frame: Screening, vaccination weeks 3, 4 and 6; 2 weeks post last vaccination and 3, 6 and 12 months post first vaccination.
Population: as for outcome 4
Measure: Mean (Full Range); unit: Fold Change from Baseline
Arm/Group | Participants With Advanced NSCLC, to Receive AST-VAC2
Number analyzed (Participants) | 8
Fold Change from Baseline
  Week 3 Vaccination: number analyzed (Participants) | 6
  Week 3 Vaccination | 43.79 [43.79 to 43.79]
  Week 4 Vaccination: number analyzed (Participants) | 5
  Week 4 Vaccination | 285.10 [32.11 to 538.00]
  Week 6 Vaccination | 515.34 [34.68 to 996.00]
  2 weeks post last vaccination: number analyzed (Participants) | 4
  2 weeks post last vaccination | 42.53 [42.53 to 42.53]
  3 months post first vaccination: number analyzed (Participants) | 4
  3 months post first vaccination | 45.68 [45.68 to 45.68]
  6 months post first vaccination: number analyzed (Participants) | 3
  6 months post first vaccination | 49.11 [49.11 to 49.11]
  12 months post first vaccination: number analyzed (Participants) | 2
  12 months post first vaccination | 88.20 [88.20 to 88.20]

7. Secondary Outcome: Tumour Response According to Immune-Related Response Criteria (irRC) Post Vaccination
Description: Number of participants with complete response, partial response, stable disease, progressive disease or who were not evaluable at radiological disease assessment (computerised tomography and/or magnetic resonance imaging) at the End of Vaccination visit according to irRC (Appendix 3 of protocol).
Time Frame: Radiological disease assessment at Baseline and End of Vaccination visit (30 days post last vaccination), up to 94 days.
Population: Response Population: All eligible participants who have received at least one AST-VAC2 vaccination and have had a baseline assessment of disease and at least one repeat disease assessment measured according to irRC. For details of irRC, refer to Appendix 3 of the study protocol. Participants with rapid tumour progression before completion of 6 AST-VAC2 vaccinations were classified as early progression and included in the Response Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Advanced NSCLC, to Receive AST-VAC2
Number analyzed (Participants) | 8
Participants
  Progressive disease (irPD) | 3
  Stable disease (irSD) | 5

8. Secondary Outcome: Overall Survival at 2 Years Post First Vaccination
Description: Number of participants alive at 2 years post their first vaccination.
Time Frame: From first AST-VAC2 vaccination to 2 years post first vaccination.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Advanced NSCLC, to Receive AST-VAC2
Number analyzed (Participants) | 8
Participants
  Alive | 3
  Deceased | 5

ADVERSE EVENTS:
Time Frame: Safety data were collected from the time of informed consent until 2 years from the first dose of AST-VAC2 for this interim report. Participants were to be followed-up for 5 years and any changes to information reported at end of trial updated. However, no participants continued beyond 2 years and end of trial was reached. Median (range) time from informed consent to end of follow-up was 402.5 days (101-770).
Description: AEs and SAEs collected until 30 days post last vaccination; only related AEs and SAEs collected thereafter. AE terms from vocabulary MedDRA v25.0. Reported for the Safety Population: all enrolled participants who received at least one AST-VAC2 vaccination (N=8). All-cause mortality reported for all participants (N=9), including those who died prior to receiving AST-VAC2 (n=1) or during survival follow-up for reasons unrelated to AST-VAC2 (n=5) and that were not part of the safety analyses.
Arm/Group | Participants With Advanced NSCLC, to Receive AST-VAC2
All-Cause Mortality (participants affected / at risk) | 6/9
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Advanced NSCLC, to Receive AST-VAC2 (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Axillary pain (General disorders) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 6 (10)
Headache (Nervous system disorders) | 1 (4)
Hot flush (Vascular disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Influenza like illness (General disorders) | 2 (2)
Infusion related hypersensitivity reaction (Immune system disorders) | 1 (1)
Injection site reaction (General disorders) | 8 (41)
Insomnia (Psychiatric disorders) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Swelling (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaccination site pain (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
An interim report presenting data for 2-year follow-up was planned as participants were to be followed-up for 5 years for safety. However, no participants continued beyond 2 years and end of trial was reached, so there will be no further data beyond the 2-year follow-up reported here.

Due to difficulties in interpretation of non-durable response versus limitations of the ELISPOT assay, only durable response has been reported for clarity for outcome measure 5.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT03371485/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT03371485/SAP_001.pdf